CLINICAL TRIAL: NCT02521883
Title: Transcranial Direct Current Stimulation (tDCS) as an add-on Therapy for Treatment of Major Depressive Disorder. (DEPTDCS2014)
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Turku University Hospital (Other Government)
Collaborators: Tampere University Hospital (Other); Sooma Oy (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: T248/2014
Record Dates: First submitted 2015-08-11; First posted 2015-08-13 (Estimated); Last update posted 2018-09-12 (Actual); Status verified 2018-09

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Device: Sooma tDCS (Active Comparator): The active group will receive active Sooma tDCS treatment for the first three weeks followed by maintenance treatments at weeks 5 and 6.
  Interventions: Device: Sooma tDCS
- Device: Sham tDCS (Placebo Comparator): The placebo group will receive sham tDCS treatment for the first three weeks followed by sham maintenance treatments at weeks 5 and 6.
  Interventions: Device: Sham tDCS

INTERVENTIONS:
Device: Sooma tDCS — 2mA current applied for 30 minutes in electrode locations F3 (anode) and F4 (cathode).
  Arms: Device: Sooma tDCS
Device: Sham tDCS — sham stimulation (current phased off after 20 secs) applied for 30 minutes in electrode locations F3 (anode) and F4 (cathode).
  Arms: Device: Sham tDCS

SUMMARY:
The aim is to investigate the safety and effectiveness of transcranial Direct Current Stimulation (tDCS) in patients with moderate to severe major depression compared to patients treated with conventional therapy. The tDCS will be used as add-on to conventional therapy.

This is a randomized 2-arm parallel, double blind study comparing 2 groups of 60 patients.

ELIGIBILITY:
Inclusion Criteria:

* Fulfils the ICD-10 diagnostic criteria for moderate or severe major depressive episode (F32), or recurrent major depressive episode (F33)
* Able to understand the purpose and potential risks of the study
* Able to sign informed consent

Exclusion Criteria:

* intracranial metal implants or other foreign intracranial metal object
* history of neurological conditions e.g. epilepsy, stroke (ischemic or haemorrhagic); brain tumor; increased intracranial pressure etc.
* schizophrenia
* bipolar disorder
* psychotic disorder
* substance abuse or dependency
* contra-indications to tDCS
* personality disorder that may prevent him/her to commit to the study
* skin lesion in the area of stimulation
* planned treatment of current depressive episode with ECT or rTMS

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2015-03; Primary Completion 2019-12 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Montgomery-Åsberg depression scale (MADRS) | baseline, wk 2, wk 4, wk 5, wk 6, 3 months, 6 months
  Efficacy

SECONDARY OUTCOMES:
Dichotomised response measured with MADRS. | baseline, wk 2, wk 4, wk 5, wk 6, 3 months, 6 months
  Response to treatment is defined as a ≥ 50% reduction in the MADRS baseline score.
Change from baseline in Beck Depression Inventory (BDI) scale. | baseline, wk 2, wk 4, wk 5, wk 6, 3 months, 6 months
Dichotomised remission measured with MADRS. | baseline, wk 2, wk 4, wk 5, wk 6, 3 months, 6 months
  Remission is defined as a MADRS score ≤ 10.

CONTACTS AND LOCATIONS:
Overall Officials: Tero Taiminen, MD, docent, Principal Investigator — Turku University Hospital
Locations (4):
- Finland (3):
  - PHSOTEY, Psykiatrian tulosalue, ECT-yksikkö, Lahti
  - VSSHP Psykiatria, Liedon aikuispsykiatrian poliklinikka, Lieto
  - Turku University Hospital, Turku
- Sektionen för affektiva sjukdomar, Norra Stockholms Psykiatri, Stockholms läns sjukvårdsområde, Stockholm, Stockholm County, Sweden